CLINICAL TRIAL: NCT06585644
Title: Furmonertinib in Combination with Anlotinib and Chemotherapy As Neoadjuvant Treatment for Resectable, Stage II-III EGFR-Mutated Non-Small Cell Lung Cancer: a Single-Arm, Open-Label, Phase II Clinical Trial
Brief Title: A Clinical Trial of Furmonertinib Combination Therapy As Neoadjuvant Treatment in Resectable EGFR-Mutated NSCLC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Haifeng Wang, Professor, Shanghai Pulmonary Hospital, Shanghai, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STAR 008
Record Dates: First submitted 2024-09-03; First posted 2024-09-05 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Lung Cancer (NSCLC)
Keywords: Neoadjuvant; EGFR-mutant non-small-cell lung cancer; Furmonertinib; Anlotinib
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — aflutinib; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment group (Experimental): Furmonertinib in combination with anlotinib and chemotherapy as a neoadjuvant treatment regimen. The enrolled patients will take furmonertinib, with a dose of 80mg/d, from day 1 to day 21, q3w/cycle; and anrotinib, with a dose of 12mg/d, from day 1 to day 14, q3w/cycle. They will receive furmonertinib and anrotinib treatment for 3 cycles, and combined platinum-based chemotherapy for 4 cycles. CT assessment (RECIST1.1) will be conducted within 3 weeks after the completion of treatment. All patients will undergo radical lung lobectomy and systemic lymph node dissection 3 weeks after the end of treatment. Patients who undergo surgery (CR+PR+SD) will take furmonertinib at a dose of 80mg/d for 1 year. PD patients will be transferred to the oncology or radiation department for comprehensive treatment.
  Interventions: Drug: Furmonertinib in combination with Anrotinib and chemotherapy

INTERVENTIONS:
Drug: Furmonertinib in combination with Anrotinib and chemotherapy — The enrolled patients are planned to receive preoperative treatment with a combination of furmonertinib and anrotinib, along with platinum-based doublet chemotherapy. Three weeks after the completion of this treatment, they will undergo curative lung lobe resection and systemic lymph node dissection. Postoperatively, they will continue taking furmonertinib for one year. In case of disease progression, they will be switched to comprehensive therapy.
  Other Names: Treatment regimen of Furmonertinib in combination with Anrotinib and chemotherapy

SUMMARY:
Evaluate the efficacy and safety of neoadjuvant furmonertinib combined with anlotinib and chemotherapy in patients with resectable stage II-III EGFR mutation-positive non-small cell lung cancer.

DETAILED DESCRIPTION:
Furmonertinib is a third-generation EGFR-TKI developed by Shanghai Allist Pharmaceuticals, capable of targeting both EGFR-sensitive mutations and the Thr790Met mutation. The FURLONG study demonstrated that, in Chinese patients with EGFR-mutant NSCLC, first-line treatment with furmonertinib showed superior PFS and better tolerability compared to the first-generation EGFR-TKI gefitinib, particularly in patients with central nervous system metastases. Anlotinib is a multi-target TKI developed by Chia Tai Tianqing Pharmaceutical, which can inhibit multiple kinases, including VEGFR, PDGFR, FGFR, and c-Kit, exhibiting anti-tumor angiogenesis and tumor growth inhibition effects. The FLALTER study showed that anlotinib combined with gefitinib significantly prolonged median PFS in treatment-naive metastatic EGFR-mutant NSCLC patients. Preliminary results from ongoing clinical trials indicate that the ORR of anlotinib combined with third-generation EGFR-TKIs in advanced NSCLC ranges from 65.20% to 96.15%. Compared to adjuvant therapy, neoadjuvant therapy for resectable NSCLC offers several potential benefits, including improved patient tolerance, early control of microscopic metastatic disease through systemic treatment, and the potential for less extensive surgical resection, leading to an increased rate of complete (R0) resection. So far, the exploration of EGFR-TKIs, including gefitinib, erlotinib, and osimertinib, in the field of neoadjuvant therapy has been undertaken. An open-label, single-arm Phase 2 study (NCT00188617) demonstrated that gefitinib is a safe and feasible option for unselected patients with Stage I NSCLC, with an ORR of 11%. Another single-arm Phase 2 study (NCT01833572) showed that neoadjuvant gefitinib is a feasible treatment for patients with Stage II-IIIA NSCLC harboring EGFR mutations, with an ORR of 54.5%, a MPR rate of 24.2%, and a median DFS of 33.5 months. The EMERGING-CTONG 1103 trial was the first randomized Phase 2 study comparing neoadjuvant erlotinib with chemotherapy in patients with locally advanced (Stage IIIA-N2) NSCLC with EGFR-sensitive mutations. The final results, with a median follow-up of 62.5 months, showed that the PFS in the neoadjuvant erlotinib group was significantly longer than in the chemotherapy group, although this did not translate into an OS benefit. Preliminary results from ongoing clinical trials with osimertinib suggest that this third-generation EGFR-TKI is generally safe and may be an effective neoadjuvant treatment option. This study aims to investigate the efficacy and safety of neoadjuvant furmonertinib combined with anlotinib and chemotherapy in resectable stage II-III EGFR-mutant NSCLC.

ELIGIBILITY:
Inclusion Criteria: 1) EGFR mutation-positive (including 19Del and 21L858R) non-small cell lung cancer (NSCLC) confirmed by biopsy; 2) Resectable stage II-III NSCLC confirmed by chest CT, PET-CT, and/or EBUS; 3) Absence of distant metastasis (including head MRI, whole-body bone scan, PET-CT, CT of liver and adrenal glands); 4) The patient exhibits good pulmonary function and is deemed suitable for surgical intervention; 5) Aged 18 and above; 6)At least one measurable tumor lesion (with a longest diameter of 10mm or more as measured by CT); 7) The ECOG score ranges from 0 to 1; 8) Women of childbearing age must undergo a pregnancy test within 7 days prior to treatment, and the result must be negative. During the trial period and for 30 days following its conclusion, reliable contraceptive measures such as intrauterine devices, oral contraceptives, and condoms should be utilized. Additionally, men of reproductive age should use condoms for contraception during the trial period and for 30 days after its completion; 9) The other major organs (liver, kidneys, hematological system, etc.) are functioning normally. Hemoglobin is ≥9.0 g/dL (or can be maintained or exceeded through treatments such as blood transfusions); the red blood cell count is ≥2.0×10^9/L; the absolute neutrophil count is ≥1.0×10^9/L; the platelet count is ≥100×10^9/L; total bilirubin levels are within the normal range; AST, ALT, and alkaline phosphatase levels are ≤2.5 times the upper limit of normal; creatinine level is ≤2.0 mg/dL; creatinine clearance rate is ≥60 ml/min; patients who have not received anticoagulant therapy should have a prothrombin time (PT) and activated partial thromboplastin time (aPTT) ≤ 1.5 times the upper limit of normal, while patients who have undergone comprehensive or intravenous anticoagulant therapy are eligible for clinical trials only if they have maintained stable anticoagulant drug dosages for at least 2 weeks and their coagulation test results fall within the target therapeutic range; 10) The patient is required to sign an informed consent form. Exclusion Criteria: 1) The patient has undergone comprehensive anti-cancer treatment for non-small cell lung cancer, including surgical intervention, local radiotherapy, cytotoxic drug therapy, and targeted drug therapy; 2) The patient had no history of any cancer other than small cell lung cancer within the 5 years prior to the trial, with the exception of in situ cervical cancer, cured basal cell carcinoma, and bladder epithelial neoplasms (including Ta and Tis); 3) The patient has any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, recent onset of angina within the past 3 months, congestive heart failure [≥ NYHA Class II], myocardial infarction (within the past 6 months), severe arrhythmia, and liver, kidney or metabolic disorders requiring drug therapy); 4) The patient is a carrier of active hepatitis B, hepatitis C, or HIV; 5) Patients with severe or newly developed gastrointestinal diseases presenting diarrhea as the primary symptom; 6) The patient is receiving treatment with a P-glycoprotein inhibitor; 7) Patients with a history of or current cardiovascular malformations; 8) Patients with a history of or currently suffering from interstitial lung disease; 9) Patients who have undergone major systemic surgery or experienced severe trauma within the three months prior to the trial; 10) Those afflicted with neurological disorders or psychiatric illnesses; 11) Patients experiencing malabsorption conditions; 12) Female patients who are pregnant or lactating; 13) Other situations where researchers deem the patient unsuitable for enrollment. Withdrawal Criteria: In the following cases, the patient will withdraw from the trial: 1) The patient himself or his legal representative requests withdrawal; 2) The investigator believes that the patient's continued participation in the study will be harmful to their health; 3) The patient has developed a severe allergic reaction to the chemotherapy drug, such as grade 3-4 exfoliative dermatitis or anaphylaxis; 4) There is any other serious adverse reaction, and the principal investigator (PI) or a PI-designated investigator deems it necessary to suspend treatment; 5) The patient's compliance is very poor; 6) The patient's β-HCG test result suggests pregnancy; 7) During the study period, the patient develops another disease. The investigator believes that the disease will significantly affect the evaluation of the patient's clinical condition and it is necessary to terminate the treatment plan; 8) The patient is found to have another malignant tumor that needs to be treated; 9) The patient is lost to follow-up; 10) The patient has taken illicit drugs or other substances judged by the investigator to be likely to cause toxicity or lead to a bias in the study results; 11) The patient dies. Patients who withdraw from the trial should have the reason for withdrawal documented in both the case report form and the patient's medical record. Follow-up should be conducted for all patients who withdraw due to adverse events or abnormal laboratory test results, until the adverse event is resolved or stabilized, and subsequent outcomes of the adverse events should be recorded. In cases where a patient dies during the course of the trial or within 28 days after its conclusion, it is incumbent upon the investigator to notify the sponsor. The cause of death must be meticulously detailed in the serious adverse event (SAE) report form and submitted to the ethics committee within 24 hours.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2030-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 Weeks
  According to RECIST 1.1, objective response rate (ORR) refers to the proportion of patients whose tumors have shrunk to a certain extent and maintained that response for a specific duration, including those with complete response (CR) and partial response (PR). Complete response is defined as the complete disappearance of all target lesions, with the shortest diameter of any pathological lymph nodes (including both target and non-target nodes) shrinking to less than 10mm. Partial response is characterized by at least a 30% reduction in the diameter of the target lesion compared to baseline levels. In this study, ORR is defined as the proportion of patients who completed neoadjuvant therapy before surgery and achieved either CR or PR based on CT evaluation three weeks after treatment.

SECONDARY OUTCOMES:
Major Pathological Response | 3 Weeks
  The Major Pathological Response (MPR) is defined as the proportion of patients, among all those who have completed treatment, with less than 10% residual primary tumor under microscopic examination with hematoxylin and eosin (HE) staining.
Complete Pathological Response | 3 Weeks
  Complete Pathological Response (CPR) is defined as the proportion of patients, among all those who have completed treatment, in whom there is no residual cancer in the primary tumor and lymph nodes under HE staining microscopy.
R0 Resection Rate | 3 Weeks
  The R0 resection rate is defined as the proportion of patients whose surgical margins are negative and there is no residual tissue visible under the microscope after the operation among all patients who have completed treatment.
Disease Free Survival | 5 years
  The disease-free survival (DFS) refers to the time from curative surgery to the time when the patient experiences recurrence or death due to disease progression.
Overall Survival | 5 years
  The overall survival (OS) is defined as the time from randomization to the occurrence of death from any cause in participants.
Treatment-Related Adverse Events | 3 Months
  Treatment-related adverse events refer to the number of adverse events related to the neoadjuvant treatment regimen assessed according to CTCAE V4.0.
Health-Related Quality of Life | 5 years
  The health-related quality of life (HRQOL) was evaluated according to the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-C30 & LC13, Version 3) for lung cancer patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No